CLINICAL TRIAL: NCT00939289
Title: Pilot Study of Concurrent Use of the SEVEN® and FreeStyle Navigator® Continuous Glucose Monitoring Systems in Adults With Type 1 Diabetes Mellitus
Brief Title: Concurrent Use of Two Continuous Glucose Monitoring Systems in Adults With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Andrew K. Balo / SVP, Clinical and Regulatory Affairs, and Quality Assurance, DexCom, Inc.
Other Study IDs: PTL-900070, Rev01
Record Dates: First submitted 2009-07-12; First posted 2009-07-14 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with T1DM: Adults (18+ years-old) diagnosed with type 1 diabetes mellitus; treated with multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Real-time continuous glucose monitoring with 2 commercially available Systems (DexCom SEVEN and Abbott Navigator)
  Other Names: DexCom SEVEN; Abbott Navigator

SUMMARY:
The purpose of this pilot study is to evaluate performance of the SEVEN System and the Navigator System when both devices are worn concurrently by subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Have been diagnosed with type 1 diabetes and are on multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy;
3. Willing not to inject insulin or wear an insulin pump infusion set within 3 inches from either Sensor site;
4. Willing to participate in an 8-hour in-clinic session on study Days 5, 10, and 15 and be willing to take 4 fingersticks per hour and have 4 blood draws per hour for the 8-hour duration of each of these in-clinic sessions;
5. Willing to take a minimum of 6 fingersticks per day during home use;
6. Willing to refrain from the use of acetaminophen during this study and for at least 24-hours prior to enrollment;
7. Willing not to schedule an magnetic resonance (MRI) scan, computed tomography (CT) scan, x-ray, for the duration of the study;
8. Able to speak, read, and write English.

Exclusion Criteria:

1. Have extensive skin changes/diseases that preclude wearing the Sensor on normal skin (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites;
2. Subjects who have a known allergy to medical-grade adhesives;
3. Are pregnant as demonstrated by a positive pregnancy test within 72 hours of insertion;
4. Have a hematocrit that is less than 30%, or greater than 55%;
5. Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study);
6. Have any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff handling venous blood samples (e.g., known history of hepatitis B or C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 1 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
CGM System(s) performance (relative to YSI and/or SMBG) evaluated by standard accuracy metrics | 15 days

SECONDARY OUTCOMES:
Documentation of all reported Adverse Device Effects, Serious Adverse Device Events, and Unanticipated Adverse Device Effects | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States

REFERENCES:
- [Result] Garg SK, Smith J, Beatson C, Lopez-Baca B, Voelmle M, Gottlieb PA. Comparison of accuracy and safety of the SEVEN and the Navigator continuous glucose monitoring systems. Diabetes Technol Ther. 2009 Feb;11(2):65-72. doi: 10.1089/dia.2008.0109. PMID 19243265
- [Derived] Garg SK, Voelmle M, Gottlieb PA. Time lag characterization of two continuous glucose monitoring systems. Diabetes Res Clin Pract. 2010 Mar;87(3):348-53. doi: 10.1016/j.diabres.2009.11.014. PMID 20022127